CLINICAL TRIAL: NCT05383482
Title: A Phase I/II Dose-Escalation and Efficacy/Safety Study of Afuresertib Plus Sintilimab Plus Chemotherapy in Patients With Selected Solid Tumors That Resistance to Prior Anti-PD-1/PD-L1 Treatment
Brief Title: Afuresertib +Sintilimab+Chemotherapy in Patients With Selected Solid Tumors That Resistance to Prior Anti-PD-1/PD-L1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laekna Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LAE202CN2101
Record Dates: First submitted 2022-04-20; First posted 2022-05-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor; NSCLC; Cervical Cancer; Endometrial Cancer; Esophageal Cancer; Gastric and Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms | interventions — afuresertib; Taxes; Docetaxel; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Afuresertib in combination with Sintilimab and Nab-paclitaxel (Experimental): Afuresertib in combination with Sintilimab and Nab-paclitaxel in patients with Endometrial Cancer and Cervical Cancer
  Interventions: Drug: Afuresertib; Drug: Nab paclitaxel; Drug: Sintilimab
- Afuresertib in combination with Sintilimab and Docetaxel (Experimental): Afuresertib in combination with Sintilimab and Docetaxel in patients with Gastric and Gastroesophageal Junction Adenocarcinoma, Non-Small Cell Lung Cancer and Esophageal Cancer
  Interventions: Drug: Afuresertib; Drug: Docetaxel; Drug: Sintilimab

INTERVENTIONS:
Drug: Afuresertib — Afuresertib 125 mg PO on days 1-5, 8-12, 15-19 or Afuresertib 125 mg QD
  Other Names: LAE002
Drug: Nab paclitaxel — Nab-paclitaxel 80 mg/M2 IV D1,8, Q3W or 100 mg/M2 IV D1,8, Q3W
  Arms: Afuresertib in combination with Sintilimab and Nab-paclitaxel
Drug: Docetaxel — Docetaxel 50 mg/M2 IV D1 Q3W or Docetaxel 60 mg/M2 IV D1 Q3W
  Arms: Afuresertib in combination with Sintilimab and Docetaxel
Drug: Sintilimab — Sintilimab 200 mg Q3W

SUMMARY:
This is a multicenter, open-label, dose-escalation and efficacy/safety Phase I/II study to assess RP2D, safety, tolerability and anti-tumor activity of Sintilimab + afuresertib + nab-paclitaxel or docetaxel administered as a combination therapy.

This study is designed to identify the MTD and recommended Phase II dose (RP2D) of afuresertib in combination with sintilimab and nab-paclitaxel or docetaxel, respectively, to characterize the PK profile of afuresertib in phase I and to evaluate clinical efficacy and safety of the combination therapy in phase II. The study population in phase II is the patients with one of the five selected cancers who resistant to the prior anti-PD-1/PL-1 treatments (as a monotherapy or in combination with other anti-cancer drugs including chemotherapy) , such as EC, GC/GEJC, EsC, CC, and NSCLC.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-escalation and efficacy/safety Phase I/II study to assess RP2D, safety, tolerability and anti-tumor activity of Sintilimab + afuresertib + nab-paclitaxel or docetaxel administered as a combination therapy. This study is designed to identify the MTD and recommended Phase II dose (RP2D) of afuresertib in combination with sintilimab and nab-paclitaxel or docetaxel, respectively, to characterize the PK profile of afuresertib in phase I and to evaluate clinical efficacy and safety of the combination therapy in phase II. The study population in phase II is the patients with one of the five selected cancers who resistant to the prior anti-PD-1/PL-1 treatments (as a monotherapy or in combination with other anti-cancer drugs including chemotherapy) , such as EC, GC/GEJC, EsC, CC, and NSCLC.

For phase I, the MTD is defined as the combination dose level with a DLT rate that is closest to the target toxicity rate (0.3). Patients in each dose level are planned to be enrolled in each cohort of size 3 and maximum to 9. Totally there would be no more than 42 cases in 2 combination groups (maximum 21 patients for each combination group). RP2D evaluation will be based on the observed safety profiles,PK ，PK was analyzed on 3-9 patients per dose of albumin-paclitaxel and docetaxel (pk Sample collection may be less than 3 if the group was discontinued due to DLT observed) . The dose escalation decision will be made based on the observed safety profiles of the tested combined doses and reviewed by the safety committee. The recommended combined dose level will be as follows based on BOIN dose escalation design.

Once the RP2D of Sintilimab + afuresertib + nab-paclitaxel or docetaxel has been established, a cohort consisting of 50-125 patients with stratifying for each cancer type (10 -25 patients for each cancer type) who resistant to anti-PD-1/PD-L1 or its combination therapy (except for CC and EC, who did not receive prior anti-PD-1/PD-L1 could be enrolled.

The preliminary anti-tumor efficacy of Sintilimab + afuresertib + nab-paclitaxel or docetaxel therapy will be assessed by the measurement of ORR, PFS, OS, DOR, DCR based on the tumor assessment in each of the five solid tumors. Patients with biomarkers, such as PTEN/PI3K/AKT alternations, will be analysed retrospectively as the subpopulations for their anti-tumor efficacy in each cancer type.

ELIGIBILITY:
Inclusion Criteria:

1. Be >=18 years of age on the day of signing the informed consent and be able to provide written informed consent for the trial.
2. Prior treatments:

   * In phase I, patients had at least 1 prior systemic anti-cancer treatment (including neoadjuvant/adjuvant therapy are qualified to be enrolled). Patients who resistant to anti-PD-1/PD-L1 are preferred.
   * In phase II, patients should meet the following 2 criteria simultaneously:

   A: resistant to anti-PD-1/PD-L1: previously received at least 6 weeks （2 cycles） anti-PD-1/PD-L1 (including neoadjuvant/adjuvant therapy) and progressed after anti-PD-1/PD-L1 or their combination therapies.

   B: received <=3 lines systematic therapy during recurrent/metastatic period.
3. Tumor diagnosis:

   * In phase I, patients had a histology confirmed diagnosis of locally advanced or metastatic solid tumors who had at least 1 prior systemic anti-cancer treatment including neoadjuvant/adjuvant therapy are qualified to be enrolled. The patients with the 5 selected cancer types below who resistant to prior anti-PD-1/PL-1 or its combination therapies will be enrolled with a higher priority.
   * In phase II, the patients have only the following diagnoses will be allowed:

     * CC: Patients with histologically confirmed metastatic, recurrent or persistent squamous cell carcinoma, adenosquamous carcinoma, adenocarcinoma of the cervix are allowed. The other histological types of cervical cancer will be excluded.
     * EC: Patients with histologically confirmed metastatic, recurrent or persistent Epithelial Endometrial Carcinoma with endometrioid, high grade serous, or clear cell carcinoma. The other histological types of endometrial cancer will be excluded.
     * EsC: Patients with histologically confirmed local advanced, recurrent or metastasis esophageal squamous cell carcinoma or Her2- adenocarcinoma.
     * NSCLC: Patients with histologically confirmed locally advanced, recurrent, or metastatic Non-Small Cell Lung Cancer (squamous cell carcinoma or adenocarcinoma, adenosquamous carcinoma), who have EGFR wild type status, KRAS wild type status and ALK- negative rearrangement status.
     * GC/GEJC: Patients with histologically confirmed locally advanced, recurrent, or metastatic Her2- gastric adenocarcinoma or gastroesophageal junction adenocarcinoma or squamous cell carcinoma allowed.
4. Biomarker test:

   * In phase I, the biomarker test with tumor sample is optional. However, blood test of cfDNA is required.
   * In phase II, if patient has prior tumor sample PTEN/PI3K/AKT gene alterations or immunohistochemistry test with a report, no further tumor sample biomarker test is needed, but the blood cfDNA test is still required in this study. Otherwise, patient should be able to provide archival or biopsy tumor samples for PTEN immunohistochemistry and PTEN/PI3K/AKT gene alterations, and/or the blood sample for PTEN/PI3K/AKT gene alterations for the cell-free DNA (cfDNA) test. The archival tumor tissue sample obtained better within 2 year from study enrollment or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated will be accepted for IHC test and gene sequencing test. Formalin-fixed, paraffin embedded tissue blocks are preferred to be sectioned on the slides.
   * Please contact sponsor if patient cannot provide archival or biopsy tumor samples.
5. Patients who are suitable for nab-paclitaxel or docetaxel judged by investigator.
6. Have measurable disease per RECIST 1.1 as assessed by local radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Patients must have an Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2.
8. Have adequate organ function as defined below. Specimens must be collected within 10 days prior to the start of study treatment.

   1. Hematological:

      Absolute neutrophil count (ANC) ≥ 1.5 × 109 /L Platelet count ≥100 × 109 /L Hemoglobin ≥ 90 g/L
      * Criteria must be met without granulocyte-colony stimulating factor, erythropoietin dependency and without packed red blood cell transfusion within last 2 weeks.
   2. Renal Creatinine ≤1.5 × upper limit of normal (ULN) OR Measured or calculated per institutional standard creatinine clearance (glomerular filtration rate can also be used in place of creatinine or creatinine clearance) ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN.
   3. Hepatic Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN.

      AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases).
   4. Coagulation International normalized ratio (INR) OR prothrombin time (PT) and Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy, as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
9. Fasting glucose ≤126 mg/dL or ≤7.0 mmol/L for patients without type 2 diabetes and ≤167 mg/dL or ≤9.3 mmol/L for patients with type 2 diabetes; OR glycosylated hemoglobin (HbA1c) ≤8%.
10. Life expectancy of 12 weeks or more based on investigator's assessment.
11. Patients have recovered from adverse events associated with chemotherapy, radiation and surgical operation as pre-treatment to Grade 1 or lower with CTCAE v5.0 excluding stable symptoms (e.g. alopecia, skin hyperpigmentation.).
12. Patients must agree to use effective contraception during the study and for at least 16 weeks after discontinuation as following:

    1. Total abstinence (if it is their preferred and usual lifestyle)
    2. An intrauterine device or hormone-releasing system
    3. A contraceptive implant
    4. An oral contraceptive (with additional barrier method) OR
    5. Have a vasectomized partner with confirmed azoospermia.
    6. Male patients must agree to use an adequate method of contraception.
13. Patient is able to swallow and retain oral medication without gastrointestinal diseases to interfere with drug absorption.

Exclusion Criteria:

1. Pregnancy or lactation. A woman of child-bearing potential, who has a positive urine pregnancy test prior to treatment. If the urine test is cannot be confirmed as negative, a serum pregnancy test will be required.
2. Prior anti-cancer treatment or any investigational agent within 28 days (or 5 half-lives, whichever is shorter) prior to the first dose of study drugs.
3. Patients that have previously received AKT or PI3 kinase pathway or mTOR inhibitors will not be enrolled.
4. Patients that discontinued prior anti PD-1/PD-L1 due to immune related AE.
5. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
6. With clinically uncontrolled pleural effusion/ascites (patients who do not need effusion drainage or have no significant increase in effusion 3 days after stopping drainage can be enrolled);
7. With a tumor compressing the surrounding important organs, compressing the superior vena cava, or invading the mediastinal great vessels, heart, etc.;
8. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
9. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
10. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, transitional cell carcinoma of urothelial cancer, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
11. History of seizure of condition that may predispose to seizure that needs anti-epileptic medications; brain arteriovenous malformation; or intracranial masses, such as schwannomas and meningiomas that are causing edema or mass effect.
12. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
13. Has severe hypersensitivity (≥Grade 3) to Sintilimab or afuresertib and/or any of their excipients.
14. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs) prior to the first dose of study treatment. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
15. Has a history of (non-infectious) pneumonitis that required steroids or has concurrent interstitial pneumonia.
16. Has an active infection requiring systemic therapy, active syphilis infection, active pulmonary tuberculosis infection，HIV-infection (i.e., HIV 1 or 2 antibody positive).
17. New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction within the past 6 months or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months.
18. Prolongation of corrected QTc interval, as corrected by the Fridericia's correction formula to greater than 450 mSec for males and 470 mSec for females: unless prolonged QTc interval due to right bundle branch block or left bundle branch block with a pacemaker.
19. Presence of uncontrolled hypertension (systolic blood pressure (BP) >160 mmHg or diastolic BP>100 mmHg). Patients with a history of hypertension are allowed, provided that BP is controlled to within these limits by anti-hypertensive treatment.
20. Has known untreated active Hepatitis B (defined as HBsAg (+) and HBV DNA ≥200 IU/mL (1000 copies/ml)) or active Hepatitis C virus infection (defined as HCV antibody positive and HCV-RNA level above the lower limit of detection).

    Note: Subjects with HBV DNA < 200 IU/ml or below the lower limit of detection are eligible. Those on active HBV therapy with viral loads under 200 IU/mL should stay on the same therapy throughout study treatment.
21. Has a known psychiatric or substance abuse disorder that would interfere with the patient's ability to cooperate with the requirements of the study.
22. Patients receiving a strong CYP3CA, OATP, BRCP substrate or inducer are not eligible. Please see protocol related section for the list of prohibited medications.
23. Has had an allogenic tissue/solid organ transplant.
24. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
25. Patient needs radiotherapy during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Phase I: Frequency and severity of Adverse Events (AEs),including incidence rate of DLTs | Through study completion for an average of 12 months
  Phase I: Findings on physical examination, ECG, vital signs, and reports of the laboratory results based on the CTCAE v5.0
Phase I: Recommended Phase II dose | about 12 months
  Phase I: Determining the RP2D of the Combination therapy for phase II
Phase II: Overall Response Rate (ORR) based on RECIST 1.1 | Change from Baseline beginning at Cycle 3 Day 1 and then every 6 weeks × 18weeks then every 9 weeks through study completion, an average of 2 years (each cycle is 21 days)
  Anti-tumor activity of Afuresertib in combination with Sintilimab and Nab-paclitaxel or Docetaxel in EC/CC/ GC/GEJC/EsC/NSCLC

SECONDARY OUTCOMES:
Phase I：Overall Response Rate (ORR) based on RECIST 1.1 | Change from Baseline beginning at Cycle 3 Day 1 and then every 6 weeks × 18weeks then every 9 weeks through study completion, an average of 1 year (each cycle is 21 days)
  Phase I: Anti-tumor activity of Afuresertib in combination with Sintilimab and Nab-paclitaxel or Docetaxel
Disease Control Rate (DCR) based on RECIST 1.1 | Change from Baseline beginning at Cycle 3 Day 1 and then every 6 weeks × 18weeks then every 9 weeks through study completion, an average of 1 year (each cycle is 21 days)
  Anti-tumor activity of Afuresertib in combination with Sintilimab and Nab-paclitaxel or Docetaxel
Duration of Response (DOR) based on RECIST 1.1 | Change from Baseline beginning at Cycle 3 Day 1 and then every 6 weeks × 18weeks then every 9 weeks through study completion, an average of 1 year (each cycle is 21 days)
  Anti-tumor activity of Afuresertib in combination with Sintilimab and Nab-paclitaxel or Docetaxel
Progression Free Survival (PFS) based on RECIST 1.1 | Change from Baseline beginning at Cycle 3 Day 1 and then every 6 weeks × 18weeks then every 9 weeks through study completion, an average of 1 year (each cycle is 21 days)
  Anti-tumor activity of Afuresertib in combination with Sintilimab and Nab-paclitaxel or Docetaxel
Assessing pharmacokinetics parameters | Assessed on Day 1, Day 15 of Cycle 1 and Day1 of Cycle 3 (each cycle is 21 days)
  Calculated from plasma concentrations of afuresertib obtained at various time points
Phase II: Overall Response Rate (ORR) based on immune-related iRECIST | Change from Baseline beginning at Cycle 3 Day 1 and then every 6 weeks × 18weeks then every 9 weeks through study completion, an average of 2 years (each cycle is 21 days)
  Anti-tumor activity of Afuresertib in combination with Sintilimab and Nab-paclitaxel or Docetaxel
Phase II: Overall Survival (OS) based on RECIST 1.1 | Change from Baseline beginning at Cycle 3 Day 1 and then every 6 weeks × 18weeks then every 9 weeks through study completion, an average of 2 years (each cycle is 21 days)
  Phase II: Anti-tumor activity of Afuresertib in combination with Sintilimab and Nab-paclitaxel or Docetaxel in EC/CC/ GC/GEJC/EsC/NSCLC

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Director, Principal Investigator — Beijing Cancer Hospital, China
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chengdu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Second University Hosital, Sichuan University, Chengdu, Sichuan